CLINICAL TRIAL: NCT01929928
Title: Sonicision Cordless Ultrasonic Dissection System in General Surgery: A Prospective Post-market Observational Study to Evaluate the Efficacy and Accuracy of a Cordless Ultrasonic Dissection System
Brief Title: Evaluation of Efficacy and Accuracy of a Cordless Ultrasonic Dissection System
Acronym: SCUD
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-12-03B
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2016-02

CONDITIONS: Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgical Patients

SUMMARY:
The purpose of this study is to test the efficacy of a new cordless ultrasonic dissection system.

DETAILED DESCRIPTION:
The Sonicision device offers the ability to achieve hemostasis and vessel dissection with a cordless system. The ultrasonic device yields coagulation and transection of vessels by conversion of electrical energy into ultrasonic vibration through a piezoelectric or magnetic transducer, which is the causation of heat induction at the jaws of the instrument through friction. The Sonicision device is able to seal vessels up to 5 mm and transection division of 10 cm segments. The Sonicision device features the following:

1. Cordless design to improve freedom and movement;
2. Simplified set up that may possibly increase operating room efficiency;
3. Dual-mode energy control to increase procedure focus;
4. Improved mobility secondary to cordless system.

Currently all devices are connected to a generator by a cable, which can lead to the cable wrapping around the device, tangle with other instruments and become inadvertently contaminated. There are several advantages with regards to utilization of a cordless device to include: improved intra-operative storage, avoidance of bundling multiple cords from various instruments that may limit instrument mobility and portability which may lead to the ability to operate with advanced surgical equipment in third world settings, trauma and surgery centers.

The study group will consist of 150 patients, male and female adults, who present with the need for general surgery in which an ultrasonic dissection device and/or a vessel sealing device will be utilized. Patients will be identified prospectively via consultation with the general surgeon. Data will be collected addressing the following variables: versatility, dissection time, vessel diameter, reliability, efficiency, tissue response, steam production, blood loss, tissue response, thermal spread, desiccation and sealing time. A tentative total of ten individual tissue specimens will be obtained by the surgeon during surgery and after the utilization of the Sonicision Cordless Ultrasonic Dissection System. The patient's histologic sample will be followed after surgery in order to determine efficacy of the vessel seal. Subsequently, the patient's information will be deidentified and the patient assigned a study number to which all further analysis will be tied. Patient participation will include time of surgery through discharge from the hospital. Study data will be collected and managed utilizing an electronic database.

ELIGIBILITY:
Inclusion Criteria:

General surgery in which an ultrasonic dissection device will be utilized Adult male and females age 18 and older

Exclusion Criteria:

Surgery involving bone Surgery involving contraceptive tubal occlusion Indication for emergency surgery Suspected inability or the inability to comply with trial procedures Employee at the investigational center, sponsor or sponsor's representative, relative or spouse of the investigator Emergency Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the division of Hepatobiliary Surgery at Carolinas Medical Center in Charlotte, NC.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-01; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Placement of Sonicision Cordless Ultrasonic Dissection Device | 1 year
  Evaluation of device placement will be measured based on vessel sealing variables: number of applications, vessel site, type of tissue to be sealed, number of seals to achieve hemostasis, number of activations, number of successful seals, number of failed seals, tissue sticking, tissue color, thermal spread and desiccation.
Efficacy of Sonicision Cordless Ultrasonic Dissection Device | 1 year
  Efficacy of device will be measured based on intra-operative and post-operative complication variables: estimated blood loss, blood transfusion, complications intra-operative and post-operative.

SECONDARY OUTCOMES:
Device Complications | 1 year
  Functional evaluation of device based on the variables: device malfunction, number of battery and generator changes during a procedure.

CONTACTS AND LOCATIONS:
Overall Officials: David A Iannitti, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States